CLINICAL TRIAL: NCT03714048
Title: International Observational Study on BLood Management for Mechanical Circulatory Support Using Extracorporeal Membrane Oxygenation (OBLEX)
Brief Title: Blood Management During ECMO for Cardiac Support
Acronym: OBLEX
Status: Completed | Type: Observational
Sponsor: St Vincent's Hospital, Sydney (Other)
Responsible Party: Principal Investigator, Hergen Buscher, Principal Investigator, St Vincent's Hospital, Sydney
Other Study IDs: HREC/18/SVH/202
Record Dates: First submitted 2018-10-16; First posted 2018-10-22 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Death, Sudden, Cardiac; HEART ARREST; Shock, Cardiogenic; Arrhythmias, Cardiac; Hemorrhage; Venous Thrombosis; Embolism; Blood Transfusion; Disseminated Intravascular Coagulation
Keywords: Extracorporeal Membrane Oxygenation; ECMO; VA-ECMO
MeSH Terms: conditions — Death, Sudden, Cardiac; Heart Arrest; Shock, Cardiogenic; Arrhythmias, Cardiac; Hemorrhage; Venous Thrombosis; Embolism; Disseminated Intravascular Coagulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Perioperative
- Cardiogenic shock minus arrest
- Cardiogenic shock plus arrest
- Preventive

SUMMARY:
Extracorporeal membrane oxygenation (ECMO) is a lifesaving procedure used to treat severe forms of heart and/or lung failure. It works by the principal of replacing the function of these organs by taking blood from the patient, provide it with oxygen outside the body and return it to the patient in one continuous circuit. Because of the evaluability of better technology, the use of ECMO has exponentially risen over the last decade. This treatment is very invasive and carries a number of risks. It is mostly used in situations where it seems likely that the patient would otherwise die and no other less invasive measure could change this. Still in large registries 50-60% of patients die which is often due to complications associated with the treatment.

One of the most important complication is caused by the activation of clotting factors during the contact with the artificial surfaces of the device. This can lead to clot formation inside the patient or the device. To counterbalance this anticoagulation is needed. Because of the consumption of clotting factors and the heparin therapy bleeding complications are also very common in ECMO.

Clinicians are challenged to balance these competing risks and are often forced to transfuse blood products to treat these conditions, which comes with additional risks for the patient. Many experienced centres have reported thromboembolic and bleeding events as the most important contributor to a poor outcome of this procedure. However, no international study combining the experience of multiple centres to compare their practice and identify risk factors which can be altered to reduce these risks.

This study has been endorsed by the international ECMONet and aims to observe the practice in up to 50 centres and 500 patients worldwide to generate the largest ever published database on this topic. It will concentrate on patients with severe heart failure and will be able to identify specific risk factors for thromboembolic and bleeding events. Some of these factors may be modifiable by change in practice and can subsequently be evaluated in clinical trials. Some of these factors may include target values for heparin therapy and infusion of clotting factors.

This study will directly improve patient management by informing clinicians which measures are associated with the best outcome and indirectly helps building trials to increase the evidence further.

DETAILED DESCRIPTION:
Background:

Extracorporeal Membrane Oxygenation (ECMO) is the most frequently used mechanical circulatory support (MCS) for severe forms of cardiogenic shock (CS) when simpler measures like inotropes and the intra-aortic balloon pump fail. Despite improvements in technology and growing clinical experience mortality among patients supported with ECMO remains above 40%. In addition to bloodstream infections and circuit-related complications, disorders of coagulation which can result in life-threatening hemorrhage, thrombosis and thromboembolic events remain the most frequent and dangerous complications.

Significant perturbations in hemostatic function are seen during extracorporeal therapies. The mechanisms of these are complex and relate to underlying pathology, blood-surface contact and pump mechanics. They are evidenced by platelet dysfunction and consumption, hyperfibrinolysis or coagulopathy secondary to disseminated intravascular coagulation (DIC).

Given the multifactorial disturbances of hemostasis that can result in hemorrhage during ECMO, standard laboratory hemostatic testing may not enable the clinician to specify the underlying cause of the bleeding. Consequently, bleeding events are typically managed with transfusion of coagulation factors guided by clinician judgment.

Anticoagulation practice itself may also determine the bleeding risk and it has been noted that practice is variable. Heparin dosage and titration as well as stopping rules are not well defined and vary vastly in the literature.

Historically, bleeding had been reported in clinical trials where high anticoagulation targets were used which contributed to excessive bleeding.

Bleeding and the utilization of blood products have frequently been described as a predictor of poor outcome in the general ICU population.

Guidelines suggesting high hemoglobin targets to optimize oxygen delivery in ECMO have subsequently been challenged to avoid potential risk associated with blood product transfusions.

Excessive transfusion of blood products, which increases the risk of complications such as transfusion-related acute lung injury (TRALI), transfusion-related circulatory overload (TACO) and transfusion-related immunomodulation (TRIM) may outweigh the potential benefit. Unnecessary exposure to procoagulant factors also increases the risk of ECMO-circuit malfunction and thromboembolic complications. These additionally lead to increased ICU and hospital length of stay, and markedly increased costs. Improvement in the management of anticoagulation and hemostatic therapy in this setting may alter outcome in ECMO.

Current knowledge is insufficient to provide high level evidence-based recommendations on anticoagulation, management of bleeding or transfusion triggers. Published literature is mostly drawn from retrospective single centre reports over different time periods, case mix, ECMO equipment and data points. In the absence of randomized controlled trials (RCT) addressing these multitude of issues, best practice should be based on multicenter cohort studies. A standardized multicenter approach is needed to observe associations between variations in practice and clinically relevant outcomes. These observations will support hypothesizes for future RCT and is crucial to propose feasible interventions.

Hypothesis:

• Bleeding, thromboembolic complications and blood product usage in ECMO for MCS

* Vary among centers providing the service
* Differ with different anticoagulation strategies
* Are dependent on diagnostic grouping and presentation category
* Are independently associated with morbidity and mortality

Design:

• An international, multicenter, observational cohort study.

Aim:

* To prospectively describe bleeding, thromboembolic complications, blood management and anticoagulation in ECMO for MCS.
* Investigate its associations with morbidity and mortality.
* Identify risk factors for bleeding, thromboembolic complications and blood product usage.
* To provide information on current standard of care for future prospective interventional trials.

Significance

The Extracorporeal Life Support Organization (ELSO) maintains a registry and reports 4297 annual adult ECMO runs worldwide in 2016. This number has more than doubled since 2012. Since this registry relies on voluntary contributions it is almost certainly only reporting a fraction of all global treatments. Using national insurance datasets McCarthy reports almost 3000 usages in the US in 2012 (ELSO registry: less than 1000 for North America). Using a similar approach Karagiannidis found almost 4500 annual runs in Germany in 2014 (ELSO registry: 921 for Europe in total during the same year). Using the Japanese Diagnosis Procedure Combination national inpatient database 5263 patients were treated in that country for cardiac support only over a period of 3 years from 2010 to 2013 (ELSO registry: less than 500 for the whole Asia-Pacific area). No global statistic of ECMO usage exists but it can be assumed that the largest registry probably underestimates the true utilisation by a factor of 5-20. This would translate into an annual number of patients treated with ECMO of around 20.000 to 100.000.

The mortality attributed to bleeding and thromboembolic complications is also unknown. Based on ELSO data Lorusso found the incidence of stroke, cerebral haemorrhage, brain death and seizures to be 7% with an associated mortality of more than 70% in patients treated with ECMO for respiratory support. Given that these patients were primarily diagnosed with a pulmonary disease and a low risk profile for cerebral complications, ECMO may be a contributor to this negative outcome which may potentially be avoidable. Other causes of bleeding and thromboembolic complications during ECMO for MCS are more frequent and reported as:

* Clots: oxygenator 8.2%
* Other clots in the ECMO system 5.6%
* Gastrointestinal haemorrhage 4.4%
* Cannulation site bleeding 17.5%
* Surgical site bleeding 19.2%
* Haemolysis 5.5%
* Disseminated intravascular coagulation (DIC) 3.5%
* Cardiac tamponade: blood 5%
* Pulmonary haemorrhage 2.8%
* Limb Ischemia 3.6%
* Compartment syndrome 1%
* Limb Fasciotomy 1.5%
* Limb Amputation 0.5% While these registry data do not allow insight into a causative correlation with mortality, bleeding and thromboembolic complications almost certainly contribute to morbidity and treatment costs.

The need for blood transfusions has been quantified to be between 1 and 4 Units per day of ECMO treatment which may further contribute to mortality and morbidity through direct and indirect transfusion related complications. Best strategies to avoid blood transfusions in ECMO have not been identified.

The costs directly related to ECMO are difficult to assess. However, so far the largest randomized trial has calculated the additional costs of patients treated with the modality at about 40.000 pounds while other observational studies measured a direct treatment related cost of 73.000 USD and 106.000 Euro. Even a conservative estimation of the annual case load would quantify the global treatment related costs at more than 1.5 billion USD. Using the same conservative approach and assuming an average ECMO treatment duration of 10 days would translate into 200.000 units of blood transfused. Given the reported direct costs of a blood transfusion of USD 265 the costs would be about 50 Million USD per annum for red blood cells alone. Indirect costs related to TRALI and other complications as well as administration costs cannot be assessed but are most likely much higher.

Specific data on blood management and anticoagulation have only been published in single centre retrospective trials. This study's targeted recruitment of 500 patients would represent by far the largest contemporary sample in this area worldwide.

ELIGIBILITY:
Inclusion Criteria:

* ECMO for mechanical circulatory support
* ECMO using a temporary device containing an oxygenator and an active blood pump.

Exclusion Criteria:

* ECMO for respiratory support only
* Age<18
* ECMO treatment outside the participating centre for >24 hours
* Previous enrolment in OBLEX during the same hospital admission
* ECMO treatment outside the intensive care unit only (e.g. theatre or angiography)
* Enrolment in other studies where a randomized intervention is targeting anticoagulation or blood management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All prospective patients who receive ECMO for cardiac support in a participating centre.
Sampling Method: Probability Sample
Enrollment: 561 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Hospital mortality | Till the end of the index hospital admission, on average 30 days
  Fraction of patients not surviving the index hospital admission

SECONDARY OUTCOMES:
ECMO free days | 28 days after the start of the treatment
  Number of days alive and not treated with ECMO during the first 28 days after the start of the treatment
ICU free days | 28 days after the start of the treatment
  Number of days alive and not treated in ICU during the first 28 days after the start of the treatment
Ventilator free days | 28 days after the start of the treatment
  Number of days alive and not treated with mechanical ventilation during the first 28 days after the start of the treatment
Anticoagulation management | For 7 days after the start of ECMO or till the end of treatment (whatever comes first)
  Parameter used to titrate anticoagulation, drug used and achieved values
Hemorrhagic complications | For 7 days after the start of ECMO or till the end of treatment (whatever comes first)
  Type, location and management of hemorrhage
Thromboembolic complications | For 7 days after the start of ECMO or till the end of treatment (whatever comes first)
  Type, location and management of thromboembolic complication

CONTACTS AND LOCATIONS:
Locations (1):
- St Vincent's Hospital, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Buscher H, Hayward C. Extracorporeal Membrane Oxygenation: An Expanding Role in Cardiovascular Care. Heart Lung Circ. 2018 Jan;27(1):3-5. doi: 10.1016/S1443-9506(17)31472-5. No abstract available. PMID 29198832
- [Result] Buscher H, Zhang D, Nair P. A pilot, randomised controlled trial of a rotational thromboelastometry-based algorithm to treat bleeding episodes in extracorporeal life support: the TEM Protocol in ECLS Study (TEMPEST). Crit Care Resusc. 2017 Oct;19(Suppl 1):29-36. PMID 29084499
- [Result] Smith M, Vukomanovic A, Brodie D, Thiagarajan R, Rycus P, Buscher H. Duration of veno-arterial extracorporeal life support (VA ECMO) and outcome: an analysis of the Extracorporeal Life Support Organization (ELSO) registry. Crit Care. 2017 Mar 6;21(1):45. doi: 10.1186/s13054-017-1633-1. PMID 28264702
- [Result] Buscher H, Vukomanovic A, Benzimra M, Okada K, Nair P. Blood and Anticoagulation Management in Extracorporeal Membrane Oxygenation for Surgical and Nonsurgical Patients: A Single-Center Retrospective Review. J Cardiothorac Vasc Anesth. 2017 Jun;31(3):869-875. doi: 10.1053/j.jvca.2016.10.015. Epub 2016 Oct 17. PMID 28082026
- [Result] Venkatesh K, Nair PS, Hoechter DJ, Buscher H. Current limitations of the assessment of haemostasis in adult extracorporeal membrane oxygenation patients and the role of point-of-care testing. Anaesth Intensive Care. 2016 Nov;44(6):669-680. doi: 10.1177/0310057X1604400601. PMID 27832552
- [Result] Nair P, Hoechter DJ, Buscher H, Venkatesh K, Whittam S, Joseph J, Jansz P. Prospective observational study of hemostatic alterations during adult extracorporeal membrane oxygenation (ECMO) using point-of-care thromboelastometry and platelet aggregometry. J Cardiothorac Vasc Anesth. 2015 Apr;29(2):288-96. doi: 10.1053/j.jvca.2014.06.006. Epub 2015 Feb 2. PMID 25655210
- [Result] Herbert DG, Buscher H, Nair P. Prolonged venovenous extracorporeal membrane oxygenation without anticoagulation: a case of Goodpasture syndrome-related pulmonary haemorrhage. Crit Care Resusc. 2014 Mar;16(1):69-72. PMID 24588439
- [Derived] Thao LTP, Buscher H, Nguyen TL, Martucci G, Gratz J, Trummer G, Schmidt M, Gautier M, Serra A, Takeda K, Pooth JS, Rahn K, Geismann F, Lubnow M, Retter A, Nair P, Vlok R, Siriwardena M, Winearls J, Walsham J, Gattas D, Aneman A, Fulcher B, Newman S, Reynolds C, Arcadipane A, Shekar K, Hodgson C, Pellegrino V, Mueller T, Brodie D, McQuilten Z; International ECMO Network (ECMONet). Liberal or restrictive transfusion for veno-arterial extracorporeal membrane oxygenation patients: a target trial emulation using the OBLEX study data. Crit Care. 2025 Aug 18;29(1):360. doi: 10.1186/s13054-025-05606-1. PMID 40826421